CLINICAL TRIAL: NCT04291937
Title: A Multicenter Expanded Access Treatment Protocol of Lurbinectedin (PM01183) in Previously Treated Small Cell Lung Cancer in the USA
Brief Title: A Multicenter Expanded Access Treatment Protocol of Lurbinectedin in Previously Treated SCLC in the USA
Status: Approved for marketing | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: LUR_EAP-001-2019
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Lurbinectedin — Powder for concentrate for solution for infusion in 4 mg vials
  Other Names: PM01183

SUMMARY:
This is an expanded access program in the USA to enable eligible patients with previously treated small cell lung cancer to access lurbinectedin treatment prior to FDA approval. Sites must apply to participate in the program. A medical doctor must assess whether the potential benefit outweighs the risk of the investigational therapy considering the program eligibility criteria and the individual patient's medical history.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent adult
* Confirmed and unresectable Small Cell Lung Cancer (SCLC)
* Patients must have received one prior chemotherapy containing line
* Adequate organ, hematological, kidney, metabolic and liver function
* Recovery from toxicities related to previous treatment(s)
* Pregnancy must be excluded, medically acceptable contraception method

Exclusion Criteria:

* Prior treatment with lurbinectedin
* Certain concomitant diseases/conditions
* Symptomatic, steroid-requiring or progressive CNS involvement.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult